CLINICAL TRIAL: NCT04280562
Title: Extended Home-use Trial of a Novel Device to Reduce Chronic Neuropathic Pain
Brief Title: Remote Participation (Within USA) Trial of Sana Pain Reliever
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Sana Health, Inc. (Unknown)
Responsible Party: Principal Investigator, David Putrino, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 18-2282
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-07

CONDITIONS: Neuropathic Pain; Chronic Pain; Pain
Keywords: Neuropathic pain; Pain; Wearable devices; Pain management; Neuromodulation
MeSH Terms: conditions — Neuralgia; Chronic Pain; Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, sham-controlled trial parallel arm study that will assess the effectiveness and patient perception of the benefit of the Sana Pain Reliever in individuals with chronic neuropathic pain.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- "Real" SPR (Experimental): Participants will receive the device which will run the "real" Sana Pain Reliever (SPR) protocol and a tablet with a mobile application to record pain levels and other questionnaires
  Interventions: Device: Sana Pain Reliever
- Sham SPR (Sham Comparator): Participants will receive the device which will run a sham SPR protocol and a tablet with a mobile application to record pain levels and other questionnaires
  Interventions: Device: Sham SPR

INTERVENTIONS:
Device: Sana Pain Reliever — Participants will receive the SPR device and a tablet with instructions of how to use the device and how to answer the questionnaires on the tablet mobile application. Each session with the device will last 16 minutes and run under the device's normal settings. The session consists of periods of light and sounds (beeps). Participants will be instructed to use the device each day at the end of the day prior to going to sleep and whenever they experience heightened pain during the day.
  Arms: "Real" SPR
Device: Sham SPR — Participants will receive the SPR device and a tablet with instructions of how to use the device and how to answer the questionnaires on the tablet mobile application. Each session with the device will last 16 minutes and run under the device's sham settings. The session consists of periods of light and sounds (beeps). Participants will be instructed to use the device each day at the end of the day prior to going to sleep and whenever they experience heightened pain during the day.
  Arms: Sham SPR

SUMMARY:
Randomized controlled trial to assess the effectiveness and patient perception of the benefit of the Sana Pain Reliever in individuals with chronic neuropathic pain.The study is fully remote with four study visits taking place over teleconferencing and the study devices mailed to the participants to use at home for 8-14 weeks.

DETAILED DESCRIPTION:
Chronic neuropathic pain (NP) is an extremely debilitating condition with few treatment options and many of which with multiple side effects. This will be a randomized, sham-controlled trial that will investigate the effectiveness of a novel wearable device called the Sana Pain Reliever (Sana PR) at reducing chronic neuropathic pain. The Sana PR is a device comprised of a Mask to be worn over the eyes with a pair of ear buds to be worn in ears. It displays light and sounds in a predetermined algorithm which runs for 16 minutes at a time. The underlying mechanism of action for the Sana PR is Audio Visual Stimulation (AVS), a form of non-pharmacological intervention that induces a brain wave response called Frequency Following Response (FFR), which has been used for both performance enhancement and symptom management. The device will be used with a compatible tablet application that will collect data from each session that the device is used. This data will be collected through user inputs of responses to several questionnaires. This will be an at-home trial and participants will be loaned the Sana Pain Reliever device and a tablet device to run the application for the duration of the study. The trial will last a total of 14 weeks and will involve four study visits, either in-person at the Abilities Research Center at Mount Sinai Hospital in New York City, or remotely using a video call. The trial includes two baseline sessions on weeks 0 and 2, 8 weeks of the at-home intervention, and post-intervention sessions at the end of weeks 10 and 14. Participants will be instructed to use the device at the end of the day prior to going to sleep as well as whenever they experience greater than typical pain during the day . Data during the at home portion of the trial will be recorded daily via the application. The application will also prompt participants to answer fortnightly weekly questionnaires and send out compliance reminders. Additionally, a series of pain, sleep and quality of life assessments will be completed by participants at both baseline visits, a post-intervention visit and a 4-week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of neuropathic pain
* Age of 18 years or older at time of consent
* Fluent in English
* Consistent medications for the last 4 weeks prior to the first baseline visit (week 0)

Exclusion Criteria:

* Diagnosis of photosensitive epilepsy
* Active ear or eye infection
* Vision impairments that affect perception of light in one or both eyes
* Deafness in one or both ears
* Severe depression (Score higher than 30 points on the Beck's Depression Inventory)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PT, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 104 participants consented, with 75 enrolled and randomized.
Period: Baseline Screening
Arm/Group | "Real" SPR | Sham SPR
Started | 34 | 41
Completed | 34 | 41
Not Completed | 0 | 0
Period: Study
Arm/Group | "Real" SPR | Sham SPR
Started | 34 | 41
Completed | 29 | 38
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Real" SPR | Sham SPR | Total
Number analyzed (Participants) | 34 | 41 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12.7) | 48.2 (15.2) | 45.4 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 7 | 16 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 26 | 32 | 58
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 23 | 25 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI)
Description: This scale was developed to assess both the quantitative and qualitative qualities of neuropathic pain (NP). It includes 12 items, assessing spontaneous pain, brief attacks of pain, provoked pain and abnormal sensations in the painful area. This is a sensitive tool for measuring changes in neuropathic pain after a therapeutic intervention. Full scale from 0-100 with higher score indicating more symptom intensity. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 47.6 (17.2) | 41 (20.5)
  Baseline 2 (Week 2) | 48.7 (17.6) | 41.5 (23.5)
  Post-assessment (Week 10) | 39.6 (21.9) | 34 (20.3)
  Follow up (Week 14) | 36.6 (21) | 39.1 (23.1)

2. Primary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Subscale 1: Burning Pain
Description: This scale was developed to assess both the quantitative and qualitative qualities of neuropathic pain (NP). This is a sensitive tool for measuring changes in neuropathic pain after a therapeutic intervention. Full subscale from 0-100 with higher score indicating more symptom intensity. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 59.1 (25.3) | 43.8 (31.8)
  Baseline 2 (Week 2) | 58.7 (27.5) | 44.7 (30.6)
  Post-assessment (Week 10) | 41.5 (28.2) | 34.4 (31.4)
  Follow up (Week 14) | 32.9 (27.9) | 44 (30.0)

3. Primary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Subscale 2: Pressing Pain
Description: This scale was developed to assess both the quantitative and qualitative qualities of neuropathic pain (NP).This is a sensitive tool for measuring changes in neuropathic pain after a therapeutic intervention. Full subscale from 0-100 with higher score indicating more symptom intensity. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 43.5 (27.4) | 36.6 (26.6)
  Baseline 2 (Week 2) | 47.1 (23.1) | 34.9 (27.3)
  Post-assessment (Week 10) | 38.8 (28.5) | 31.0 (27.8)
  Follow up (Week 14) | 31.9 (30) | 35.0 (24.7)

4. Primary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Subscale 3: Paroxysmal Pain
Description: as for outcome 2
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 53.6 (26.9) | 42.2 (31.3)
  Baseline 2 (Week 2) | 52.9 (26.4) | 42.5 (30.8)
  Post-assessment (Week 10) | 42.5 (31.0) | 30.7 (30.5)
  Follow up (Week 14) | 43.8 (28.1) | 41.4 (31.9)

5. Primary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Subscale 4: Evoked Pain
Description: as for outcome 2
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 36.4 (24.6) | 35.2 (26.1)
  Baseline 2 (Week 2) | 39.5 (29.5) | 39.4 (28.7)
  Post-assessment (Week 10) | 33.5 (27.8) | 30.3 (25.2)
  Follow up (Week 14) | 29.7 (28.2) | 32.8 (28.9)

6. Primary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Subscale 5: Paresthesia or Dysesthesia
Description: This scale was developed to assess both the quantitative and qualitative qualities of neuropathic pain (NP). It includes 12 items, assessing spontaneous pain, brief attacks of pain, provoked pain and abnormal sensations in the painful area. This is a sensitive tool for measuring changes in neuropathic pain after a therapeutic intervention. Subscale from 0-100. Full scale from 0-100 with higher score indicating more symptom intensity. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 56.8 (26.7) | 51.2 (30.8)
  Baseline 2 (Week 2) | 54.8 (26.5) | 48.8 (32.1)
  Post-assessment (Week 10) | 45.6 (28.8) | 45.6 (28.8)
  Follow up (Week 14) | 46.3 (30.0) | 48.2 (30.1)

7. Secondary Outcome: Change in Patient Health Questionnaire Type 9 for Depression (PHQ-9)
Description: The Questionnaire Type 9 for Depression (PHQ-9) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care and is used to monitor the severity of depression and response to treatment. Full scale from 0-27, with higher score indicating more severe symptoms. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 5.8 (3.2) | 5.6 (4.5)
  baseline 2 (Week 2) | 7.4 (3.9) | 6.1 (4.5)
  Post-assessment (Week 10) | 5.9 (6.1) | 5.5 (4.6)
  Follow Up (Week 14) | 6.4 (5.2) | 6.0 (5.1)

8. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. Full score from 0-21, with higher score indicating worse sleep quality. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 9.1 (3.8) | 10.3 (3.8)
  baseline 2 (Week 2) | 9.0 (3.7) | 10.1 (4.3)
  Post-assessment (Week 10) | 7.4 (4.7) | 8.0 (5.0)
  Follow up (Week 14) | 8.7 (4.4) | 9.2 (4.1)

9. Secondary Outcome: Change in Beck Depression Inventory (BDI)
Description: The Beck Depression Inventory (BDI) is used to evaluate depression symptoms, which are estimated to be highly prevalent in chronic pain populations. This questionnaire is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Depression may be a major contributor to a lack of reduction of pain. Scoring is from 0 (minimal) to 3 (severe), with total score from 0-63. Higher total scores indicate more severe depressive symptoms. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 8.6 (6.0) | 8.0 (5.4)
  baseline 2 (Week 2) | 10.0 (7.3) | 10.0 (7.3)
  Post-assessment (Week 10) | 8.8 (7.7) | 8.3 (6.4)
  Follow Up (Week 14) | 8.6 (7.0) | 9.0 (7.2)

10. Secondary Outcome: Change in General Anxiety Disorder 7-item Questionnaire (GAD-7)
Description: The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). The items that users are asked to rank levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more symptoms. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 6.4 (4.2) | 5.0 (3.8)
  baseline 2 (Week 2) | 6.3 (3.3) | 5.7 (4.5)
  Post-assessment (Week 10) | 6.0 (5.2) | 3.9 (3.4)
  Follow up (Week 14) | 5.8 (4.3) | 4.0 (3.6)

11. Secondary Outcome: Change in World Health Organization Quality of Life Pain (WHOQOL-pain) - Pain Facet
Description: The WHOQOL-pain scale is for a specific focus on the impact of pain on QOL. The WHOQOL-pain has 22 items on the pain and discomfort module (PDM) and the importance of items within a user's daily life. The Pain facet has 4 items (1-5) which are averaged to produce the WHOQOL-Pain Pain Facet. Full scale from 1-5 with higher score indicating higher quality of life. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 2.6 (0.5) | 2.7 (0.5)
  baseline 2 (Week 2) | 2.7 (0.5) | 2.7 (0.6)
  Post-assessment (Week 10) | 2.9 (0.7) | 3.2 (0.7)
  Follow up (Week 14) | 2.9 (0.8) | 3.0 (0.7)

12. Secondary Outcome: Change in World Health Organization Quality of Life Bref (WHOQOL-BREF)
Description: The WHOQOL-BREF is a used to produce a quality of life profile for an individual that is derived from four domains. There are 26 questions which ask users to respond to quality of life (QOL) questions on a scale of 1-5 (1-Not at All, Very Poor, or Very Dissatisfied; 5- Completely, Very Good, or Very Satisfied). The QOL domain assess quality of life and has a score from 1-100. Full scale from 0-100 with higher score indicating higher quality of life. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Time Frame: Baseline 1(Week0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  baseline 1 (Week 0) | 50.4 (21.0) | 54.6 (21.8)
  baseline 2 (Week 2) | 51.8 (23.2) | 50.9 (22.6)
  Post-assessment (Week 10) | 57.7 (24.2) | 59.0 (22.7)
  Follow up (Week 14) | 50.5 (21.3) | 52.1 (22.4)

13. Secondary Outcome: Change in Patient's Global Impression of Change (PGIC)
Description: The Patient's Global Impression of Change (PGIC) will be used to assess self-reported relieving effect. It will evaluate pain from no change (score 0-1), minimally improved (score 2-3), much improved (score 4-5), and very much improved (score 6-7). The patients will answer the following question: "Since beginning treatment at this program, how would you describe the change (if any) in activity limitations, symptoms, emotions, and overall quality of life related to your condition?". Full score from 0-7, with higher score indicating more improvement. Change in score at Week 14 as compared to Week 10.
Time Frame: Post-assessment (Week 10); Follow up (Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  Post-assessment (Week 10) | 2.8 (1.9) | 2.9 (1.9)
  Follow up (Week 14) | 2.7 (1.9) | 2.5 (2.1)

14. Secondary Outcome: Visual Analogue Scale (VAS)-Pain
Description: Visual Analog Scale (VAS) to measure pain: a measure of "no pain" to "Worst pain imaginable" along a line. Participants will be asked to mark the level of their pain along the line. Full scale from 0-100 with higher score indicating more pain.
Time Frame: before and after each time device used up to 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
score on a scale
  before device use | 64.4 (17.5) | 55.9 (25.6)
  after device use | 49.6 (23.8) | 52.1 (26.9)

15. Secondary Outcome: Visual Analogue Scale (VAS)-Sleep
Description: Visual Analog Scale (VAS) to measure sleep: a measure of "did not sleep at all" to "best possible night's sleep" along a line. Participants will be asked to mark the level of their sleep along the line. The Sana Health application will prompt users to answer this scale before they use the device for the first time each day. A linear mixed model used the daily sleep-vas scores to estimate the percent of change for both arms over the course of the study (Baseline to Week-14). Percent change from mean of first 3 days. 1% to 100% with higher score indicating improved sleep quality.
Time Frame: first 3 days and 14 weeks
Measure: Mean (Standard Error); unit: percent change
Arm/Group | "Real" SPR | Sham SPR
Number analyzed (Participants) | 34 | 41
percent change | 15.7 (1.7) | 6.26 (2.5)

ADVERSE EVENTS:
Time Frame: 14 Weeks
Arm/Group | "Real" SPR | Sham SPR
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/41
Other Adverse Events (participants affected / at risk) | 4/34 | 1/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | "Real" SPR (N=34) | Sham SPR (N=41)
Neuropathic Pain Event or Increase (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT04280562/Prot_SAP_002.pdf
  • Informed Consent Form (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT04280562/ICF_001.pdf